CLINICAL TRIAL: NCT02046395
Title: Effect of Renin-angiotensin-system Blockade on Urinary Free Light Chains in Patients With Type 2 Diabetes Mellitus
Acronym: UFLC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 258683
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes; Hypertension
Keywords: Type 2 Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Amlodipine; Hydralazine; Terazosin; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Washout Period for 30 days (Other): In the washout period, the Ace Inh or ARB classes of medicine(s) that are part of the patient's antihypertensive regimen will be discontinued. The patient will be started on alternative therapy with medications that are approved by the Food and Drug Administration for treatment of high blood pressure (such as amlodipine, hydralazine, terazosin or Hydrochlorothiazide) for control of their blood pressure. The goal for their blood pressure will be set at < 140/90 mm/Hg. The washout period will last for four weeks at the end of which the patient will enter the test period.
  Interventions: Drug: amlodipine, hydralazine, terazosin or hydrochlorothiazide

INTERVENTIONS:
Drug: amlodipine, hydralazine, terazosin or hydrochlorothiazide — In the washout period, the Ace Inh or ARB classes of medicine(s) that are part of the patient's antihypertensive regimen will be discontinued. The patient will be started on alternative therapy with medications that are approved by the Food and Drug Administration for treatment of high blood pressure (such as amlodipine, hydralazine, terazosin or Hydrochlorothiazide) for control of their blood pressure.
  Other Names: Norvasc

SUMMARY:
The purpose of this study is to study the effect of blocking the renin angiotensin system on urinary free light chain excretion as compared to urine microalbumin creatinine ratio in subjects with type 2 diabetes. The long term goal is to assess urinary free-light chains as a biomarker of earlier detection of kidney function impairment in subjects with diabetes mellitus.

DETAILED DESCRIPTION:
Free light chains (FLCs) are low-molecular-mass molecules (kappa and lambda light chains), which are by-products of normal immunoglobulin synthesis and are normally excreted through the kidneys. Presence of light chains in the urine is a marker of tubular dysfunction. In patients with impaired kidney function, serum concentrations and urinary excretion of polyclonal FLCs have been noted to be increased. Increased excretion of FLCs and other low-molecular weight proteins [cystatin C, NGAL] in the urine may contribute to progression of chronic kidney disease. Higher Cystatin C has been demonstrated to be related to development of albuminuria. Neutrophil gelatinase-associated lipcalin (NGAL) excretion in the urine is a marker of tubular injury in the kidney and has been shown to be elevated in subjects with type 1 and 2 diabetes mellitus (DM). Angiotensin-converting enzyme inhibitors (Ace Inh) and angiotensin II receptor blockers (ARB) class of drugs are renoprotective in nature and are the first line therapy for treatment of diabetic nephropathy. There is no longitudinal data evaluating the effect of Ace Inh and ARB class of drugs on urinary FLCs (UFLCs).

Our hypothesis is that UFLCs are increased in patients with DM with and without kidney disease and that treatment with Ace Inh and/or ARB will decrease UFLCs in these patients. Additionally, we will explore the change in other low molecular weight proteins [cystatin C, and NGAL] in response to treatment with Ace Inh and ARB.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Hypertension
* Estimated glomerular filtration rate (eGFR) > 30 ml/min
* Use of Ace Inh and ARB for control of blood pressure who are willing to be placed on alternate drug(s) in the washout period for blood pressure control

Exclusion Criteria:

* Pregnancy
* Patients with chronic kidney disease stage with eGFR < 30 ml/min (CKD stage IV and V)
* Nephrotic range proteinuria (urinary protein > 3.5 gm/day)
* History or renal transplantation
* History of multiple myeloma
* Known history of hypersensitivity reaction or intolerability to Ace Inh or ARB.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vechi Batuman, MD, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Tulane University Health Sciences Center, New Orleans, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Alternate Antihypertensive Arm: In the washout period, the Ace Inh or ARB classes of medicine(s) that are part of the patient's antihypertensive regimen will be discontinued. The patient will be started on alternative therapy with medications that are approved by the Food and Drug Administration for treatment of high blood pressure (such as amlodipine, hydralazine, terazosin or Hydrochlorothiazide) for control of their blood pressure. The goal for their blood pressure will be set at < 140/90 mm/Hg. The washout period will last for four weeks at the end of which the patient will enter the test period.
  amlodipine, hydralazine, terazosin or hydrochlorothiazide: In the washout period, the Ace Inh or ARB classes of medicine(s) that are part of the patient's antihypertensive regimen will be discontinued. The patient will be started on alternative therapy with medications that are approved by the Food and Drug Administration for treatment of high blood pressure (such as amlodipine, hydralazine, terazosin or Hydrochlorothiazide) for control of their blood pressure.
Period: Pre RAS Blockade Washout Period
Arm/Group | Alternate Antihypertensive Arm
Started | 28
Completed | 28
Not Completed | 0
Period: RAS Blockade Washout Period
Arm/Group | Alternate Antihypertensive Arm
Started | 28
Completed | 28
Not Completed | 0
Period: Post RAS Blockade Washout Period
Arm/Group | Alternate Antihypertensive Arm
Started | 28
Completed | 27
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alternate Antihypertensive Arm
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.61 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.01 (0.23)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 72.44 (21.8)
Hemoglobin A1c [Mean (Standard Deviation); unit: Percent] | 7.53 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Change in Urine Microalbumin Creatinine Ratio
Description: Kidney function will be assessed throughout the study to assess changes in function prior to the washout of ACE/ARB medication and reintroduction of the ACE/ARB medication.
Time Frame: Visit 1 (Baseline), Visit 3 (Day 60)
Population: Measurement was done for the change between Visit 1 (screening visit and the beginning of the washout period may be combined -day -30), and Visit 3 (day 30 of the test period).
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Alternate Antihypertensive Arm
Number analyzed (Participants) | 28
mg/g | 15 (2.5)

2. Secondary Outcome: Change in the Level of Urinary Free Light Chains
Description: In relation to kidney function and washout/reintroduction of ACE/ARB medication the level of urinary free light chains will be assessed.
Time Frame: Visit 1 (Baseline), Visit 3 (Day 60)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Alternate Antihypertensive Arm
Number analyzed (Participants) | 28
mg/g | 1.14 (2.03)

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Alternate Antihypertensive (Pre RAS Blockade Washout Period): Patients underwent screening visits and continued their original antihypertensive regimens before they entered the washout period.
- Alternate Antihypertensive (RAS Blockade Washout Period): In the washout period, the Ace Inh or ARB classes of medicine(s) that are part of the patient's antihypertensive regimen will be discontinued. The patient will be started on alternative therapy with medications that are approved by the Food and Drug Administration for treatment of high blood pressure (such as amlodipine, hydralazine, terazosin or Hydrochlorothiazide) for control of their blood pressure. The goal for their blood pressure will be set at < 140/90 mm/Hg. The washout period will last for four weeks at the end of which the patient will enter the test period.
  amlodipine, hydralazine, terazosin or hydrochlorothiazide: In the washout period, the Ace Inh or ARB classes of medicine(s) that are part of the patient's antihypertensive regimen will be discontinued. The patient will be started on alternative therapy with medications that are approved by the Food and Drug Administration for treatment of high blood pressure (such as amlodipine, hydralazine, terazosin or Hydrochlorothiazide) for control of their blood pressure.
- Alternate Antihypertensive (Post RAS Blockade Washout Period): Patients were restarted on their original antihypertensive medication which they were taking when they entered the study
Arm/Group | Alternate Antihypertensive (Pre RAS Blockade Washout Period) | Alternate Antihypertensive (RAS Blockade Washout Period) | Alternate Antihypertensive (Post RAS Blockade Washout Period)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-07-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT02046395/Prot_SAP_000.pdf